CLINICAL TRIAL: NCT06150716
Title: A Phase 1b Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of Intrathecally Administered ION356 in Patients With Pelizaeus Merzbacher Disease
Brief Title: Orbit Study: A Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Intrathecally Administered ION356 in Participants With Pelizaeus Merzbacher Disease (PMD)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ION356-CS1; 2022-502432-39 (EudraCT Number)
Record Dates: First submitted 2023-11-21; First posted 2023-11-29 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Pelizaeus-Merzbacher Disease
MeSH Terms: conditions — Pelizaeus-Merzbacher Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: ION356 Dose A (Experimental): Participants will receive ION356 intrathecally at Dose A in the MAD Period, followed by ION356 Dose A in the LTE Period.
  Interventions: Drug: ION356
- Cohort B: ION356 Dose B (Experimental): Participants will receive ION356 intrathecally at Dose B in the MAD Period, followed by ION356 Dose B in the LTE Period.
  Interventions: Drug: ION356

INTERVENTIONS:
Drug: ION356 — Administered as intrathecal (IT) injection.

SUMMARY:
The primary purpose of this study is to evaluate the safety and tolerability of ION356.

DETAILED DESCRIPTION:
This is a Phase 1b, open-label multiple-ascending dose (MAD) study of ION356 in approximately 24 pediatric participants with Pelizaeus-Merzbacher Disease and genetic confirmation of proteolipid protein 1 (PLP1) gene duplication. The study will have 2 parts: a 48-week multiple-ascending dose (MAD) part followed by a long-term extension (LTE) part of 109 weeks. Eligible participants will receive doses of ION356 during the MAD portion of the study and upon completion will seamlessly transition to the open-label LTE to receive doses of ION356.

ELIGIBILITY:
Key Inclusion Criteria

1. Participant's parent or legally accepted representative can provide informed consent, attend all scheduled study visits, provide feedback regarding the participant's symptoms, and can comply with all study requirements.
2. Diagnosis of PMD with genetic confirmation of PLP1 gene duplication.
3. Clinical phenotype and brain imaging consistent with a diagnosis of PMD.
4. Male between the ages of 2 and 17 years, inclusive, at the time of informed consent.
5. Able and willing to meet all study requirements (in the opinion of the Investigator), including travel to Study Center, procedures, measurements, and visits.

Exclusion Criteria

1. Clinically significant abnormalities in medical history, laboratory tests or physical examination.
2. Unwillingness to comply with study procedures, including follow-up, as specified by this protocol, or unwillingness to cooperate fully with the Investigator.
3. Any contraindication or unwillingness to undergo magnetic resonance imaging (MRI).
4. Treatment with another investigational drug, biological agent, or device within 1 month of Screening, or 5 half-lives of the investigational agent, whichever is longer.
5. Previous treatment with an oligonucleotide (including small interfering ribonucleic acid) within 4 months of Screening if a single dose was received, or within 12 months of Screening if multiple doses were received. This exclusion does not apply to vaccines (both messenger ribonucleic acid [mRNA] and viral vector vaccines).
6. History of gene therapy or cell transplantation, or any experimental brain surgery.
7. Current obstructive hydrocephalus.
8. Known brain or spinal disease or previous spinal surgery that would interfere with the lumbar puncture (LP) process, CSF circulation, or safety assessment.
9. Hospitalization for any major medical or surgical procedure involving general anesthesia within 12 weeks prior to Screening or planned during the study.
10. Have any other conditions, which, in the opinion of the Investigator, would make the participant unsuitable for inclusion, or could interfere with the participant participating in or completing the study.

Ages: 2 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Only males are included for this disease condition.
Enrollment: 24 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs | Up to Week 145
Number of Participants With Clinically Significant Change from Baseline in Laboratory Assessments | Baseline up to Week 145
Number of Participants With Clinically Significant Change From Baseline in Neurological Examination Findings | Baseline up to Week 145
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline up to Week 145
Number of Participants With Clinically Significant Change From Baseline in Electrocardiography (ECG) | Baseline up to Week 145
Number of Participants With Change From Baseline in Concomitant Medication Use | Baseline up to Week 145

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of ION356 | Pre-dose and at multiple points post-dose up to Week 145
Area Under the Concentration-time Curve (AUC) of ION356 | Pre-dose and at multiple points post-dose up to Week 145
Plasma Terminal Elimination Half-life (t½) of ION356 | Pre-dose and at multiple points post-dose up to Week 145
Plasma Concentration of ION356 | Pre-dose and at multiple points post-dose up to Week 145
Cerebrospinal Fluid (CSF) Concentration of ION356 | Pre-dose and at multiple points post-dose up to Week 105
Concentration of ION356 Excreted in Urine | Pre-dose and at multiple points post-dose on Week 1 and Week 49
Percent of ION356 Dose Excreted in Urine | Pre-dose and at multiple points post-dose on Week 1 and Week 49
Renal Clearance of ION356 | Pre-dose and at multiple points post-dose on Week 1 and Week 49

CONTACTS AND LOCATIONS:
Locations (7):
- United States (3):
  - Ionis Investigative Site, Atlanta, Georgia
  - Ionis Investigative Site, Philadelphia, Pennsylvania
  - Ionis Investigative Site, Salt Lake City, Utah
- Ionis Investigative Site, Le Kremlin-Bicêtre, France
- Ionis Investigative Site, Göttingen, Germany
- Ionis Investigative Site, Tokyo, Japan
- Ionis Investigative Site, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Ionis may share anonymized individual participant data, aggregated clinical data, and other types of data that support the results in this study. Data requests from qualified researchers will be considered once all three of the following criteria are met: (1) 12 months from marketing approval of the study drug in both the United States and European Union; (2) 18 months from conclusion of the study; and (3) 6 months from publication of study article. Access would be via a secure environment and is contingent upon approval of a research proposal and entry into an appropriate data use agreement. Requests to access data can be submitted via the website https://vivli.org/ourmember/ionis/.